CLINICAL TRIAL: NCT00962494
Title: Cancer Survivors Online Self-Management Workshop
Brief Title: Cancer: Thriving and Surviving Online Workshop and Study for Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Hawaii Cancer Research Center (Other)
Responsible Party: Principal Investigator, Kate Lorig, Professor of Medicine, Emerita, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VAR0044; SU-07292009-3460 (Other: Stanford University)
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Blood Cancer; Breast Cancer; Prostatic Neoplasms; Colorectal Neoplasms; Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Neoplasms

ARMS (1):
- online workshop (Experimental)
  Interventions: Behavioral: Cancer: Thriving and Surviving Online Workshop

INTERVENTIONS:
Behavioral: Cancer: Thriving and Surviving Online Workshop

SUMMARY:
Cancer: Surviving and Thriving is a 6-week workshop for cancer survivors. The overall goal of the study is to determine whether an online cancer survivor education and support workshop can have lasting beneficial effects in helping survivors improve their self-management of health skills and quality of life.

DETAILED DESCRIPTION:
This workshop is aimed at helping you better manage your own health and the demands placed on you because of your cancer diagnosis. It is hoped that the workshop will give you the skills needed to reduce stress and improve your quality of life. If successful, the workshop can be made available to other cancer survivors.

Each workshop is 6 weeks with new lessons each week. You will be asked to log on at your convenience 2-3 times each week for a total of 1-2 hours, to read the lessons, complete assignments, and share your ideas and experiences with your classmates. There are no requirements that participants log in at the same time.

With the moderators and other workshop participants, you will discuss:

* Healthy eating
* Managing fatigue
* Managing stress
* Starting and maintaining an appropriate physical activity program
* Getting a good night's sleep
* Dealing with difficult emotions
* Solving the problems caused by having had cancer
* Communicating better with your health care professionals
* Communicating better with your friends, family and coworkers

ELIGIBILITY:
Inclusion Criteria:Any adult (19 and over) cancer survivor living in the United States who: 1) was diagnosed within the past 5 years with a new or recurring cancer since the original diagnosis; 2) has completed their cancer treatment (surgery, radiation and/or chemotherapy); 3) isn't currently being treated for cancer except for hormonal therapy; and 4) has and email account and access to high speed internet connection. Exclusion Criteria:Not meeting the inclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Document patterns of health care utilization | 2011
Quality of Life | baseline and 6 months
Outcome Measure: Better Interactions with Oncologists | baseline and 6 months
Health Behaviors | baseline and 6 months

SECONDARY OUTCOMES:
Satisfaction with intervention | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (2):
- Stanford University School of Medicine, Stanford, California, United States
- Macmillan Cancer Support, London, UK, United Kingdom

REFERENCES:
- [Derived] Bantum EO, Albright CL, White KK, Berenberg JL, Layi G, Ritter PL, Laurent D, Plant K, Lorig K. Surviving and thriving with cancer using a Web-based health behavior change intervention: randomized controlled trial. J Med Internet Res. 2014 Feb 24;16(2):e54. doi: 10.2196/jmir.3020. PMID 24566820